CLINICAL TRIAL: NCT02629757
Title: A Study on β-elemene as Maintain Treatment for Complete Remission Patients of Newly Diagnosed Malignant Gliomas Following Standard Treatment
Brief Title: A Study on β-elemene as Maintain Treatment for Newly Diagnosed Malignant Gliomas
Acronym: β-elemene
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Zhongping Chen, Professor, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CSNO2015001
Record Dates: First submitted 2015-12-10; First posted 2015-12-14 (Estimated); Last update posted 2018-02-23 (Actual); Status verified 2018-02

CONDITIONS: Anaplastic Oligoastrocytoma; Anaplastic Astrocytoma; Glioblastoma
Keywords: High-grade glioma; chemotherapy; β-elemene
MeSH Terms: conditions — Astrocytoma; Glioblastoma; Glioma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- β-elemene (Experimental): β-elemene 600mg/d,ivdrip,d1-14,every 28 days for 1 cycle, totally 6 cycles.
  Interventions: Drug: β-elemene

INTERVENTIONS:
Drug: β-elemene — β-elemene 600mg/d,ivdrip,d1-14,every 28 days for 1 cycle, totally 6 cycles

SUMMARY:
This study is being conducted to help determine whether β-elemene as maintain treatment for complete remission patients of newly diagnosed malignant gliomas following standard treatment, is able to delay tumor growth, or impact how long people with newly diagnosed high-grade glioma.

DETAILED DESCRIPTION:
This study is being conducted to help determine whether β-elemene as maintain treatment for complete remission patients of newly diagnosed malignant gliomas following standard treatment, is able to delay tumor growth, or impact how long people with newly diagnosed high-grade glioma. β-elemene will be given 600mg/d,d1-14,q28 days for 6 cycles.

ELIGIBILITY:
Inclusion Criteria:

* - Page 3 of 4 [DRAFT] - Arms Assigned Interventions

  * Temodar Experimental: temozolomide +α-IFN Four weeks after radiotherapy, patients will be received 6 cycle of temozolomide plus α-IFN α-IFN： 3mIU (3million) Day1,3,5 of each 28 day TMZ：150 mg/m^2 daily on Days 2-6 of each 28 day study cycle and 200 mg/m^2 daily of subsequent cycles Drug: Temozolomide dosed at 200 mg/m2 (150 mg/m2 for the first cycle) daily for 5 consecutive days, repeated every 28 days

Other Names:

• Temodar Drug: α-IFN 3mIU (3million) D1，3，5

Other Names:

Minimum Age: 18 Years Maximum Age: 75 Years Gender: Both Accepts Healthy Volunteers?: No

Criteria: Inclusion Criteria:

* Age: 18 years to 75 years
* complete remission patients of newly diagnosed WHO III-IV glioma following standard treatment
* Karnofsky Performance Score ≥ 60
* Adequate bone marrow, liver and renal function
* Ability of subject to understand character and individual consequences of the clinical trial
* Written informed consent
* anticipating survival ≥2 months

Exclusion Criteria:

* Refusal to participate the study
* Known hypersensitivity or contraindication to temozolomide
* Incompletely radiation
* Pregnant or lactating females
* Malignant tumor other than brain tumor
* Contraindicated for MRI examination
* Unable to comply with the follow-up studies of this trial
* Purulent and chronic infected wounds
* Uncontrolled psychotic disorders or epilepsy
* progression disease

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2015-04; Primary Completion 2020-04 (Estimated); Study Completion 2023-05 (Estimated)

PRIMARY OUTCOMES:
Over-all survival | 5-year

SECONDARY OUTCOMES:
Quality of life | 5-year

CONTACTS AND LOCATIONS:
Overall Officials: Zhong-ping CHEN, Principal Investigator — Sun Yat-sen University
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided